CLINICAL TRIAL: NCT00068835
Title: Remediation in Developmental Dyslexia
Brief Title: Using fMRI to Evaluate Instructional Programs for Children With Developmental Dyslexia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: 5R01HD037890 (NIH)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-11

CONDITIONS: Developmental Dyslexia
Keywords: Reading; Brain imaging
MeSH Terms: conditions — Dyslexia

INTERVENTIONS:
Behavioral: Lindamood-Bell training for dyslexia

SUMMARY:
Dyslexia is a common reading disorder. Specialized instructional programs can improve reading ability in children with dyslexia. This study will use functional magnetic resonance imaging (fMRI) to examine changes in the brains of children who have taken part in these programs.

DETAILED DESCRIPTION:
Reading is a uniquely human endeavor and failure to develop this skill can lead to serious educational and emotional consequences. Reading more slowly or less accurately, as is the case in developmental dyslexia, occurs in between 5% and 15% of individuals in the United States. Developmental dyslexia significantly interferes with academic achievement and with activities of daily living that require reading skills. Although dyslexia is considered a reading disorder, dyslexia's clinical signs are varied and include deficits in the sensory domain, abnormal phonological awareness, and problems in related linguistic skills. Phonological awareness training and visual perceptual training can improve reading ability in children with dyslexia. Recent functional imaging studies on sensory and language processing in dyslexia have demonstrated involvement of the posterior temporal and inferior parietal cortical systems of the brain. However, how these brain areas are changed as a result of dyslexia treatment has not been determined.

This study will investigate the neurophysiologic changes before and after treatment in 11- to 14-year-old children immersed in Lindamood-Bell training utilizing either phonological (LiPS) or visual (Seeing Stars) strategies. These training programs have successful behavioral outcomes, but neurophysiologic changes have not been evaluated. The study will determine whether behavioral changes in reading skills result in physiological differences in the brain identifiable with functional brain imaging and whether initial physiological observations are indicative of the degree of success of the intervention.

Participant will be randomized to receive either Lindamood-Bell training, a math intervention (active control), or no intervention (passive control). The intervention will last 6 weeks; children will have both pre- and post-intervention behavioral testing and fMRI scans.

ELIGIBILITY:
Inclusion Criteria

* Developmental dyslexia diagnosis
* English speaking
* Right-handed
* General good health

Exclusion Criteria

* Metal implant, braces, or other device that prevents child from undergoing fMRI

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160
Dates: Start 2000-06; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Guinevere F. Eden, Ph.D., Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States